CLINICAL TRIAL: NCT02743169
Title: Spatial Analysis Optimization of Prehospital Services in Karachi, Pakistan to Improve Ambulance Response Times
Brief Title: Improvement of Ambulance Response Times in Karachi, Pakistan
Status: Withdrawn | Type: Observational
Why Stopped: Could not acquire data
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00085859
Record Dates: First submitted 2016-04-13; First posted 2016-04-19 (Estimated); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Emergencies
Keywords: Geographic Information Systems; Spatial Analysis; Emergency Medical Services
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard Practice: This group will consist of ambulance calls under the standard practice of Aman Foundation for ambulance placement.
- Post-Intervention: This group will consist of ambulance calls after the spatially-optimized placement of ambulances.
  Interventions: Other: Spatially-Optimized

INTERVENTIONS:
Other: Spatially-Optimized — Spatial analysis of retrospective data will be used to optimize the placement of ambulances to decrease response time from the time the call is received until the time the ambulance arrives at the patient's location.
  Groups: Post-Intervention

SUMMARY:
The investigators hypothesize that spatial analysis of the location data of ambulance calls can improve prehospital care provided by Aman Foundation in Karachi, Pakistan by decreasing ambulance response times for high acuity patients. In Aim 1, the investigators will develop a conceptual framework for prehospital care in low- and middle-income countries (LMICs) to anchor this project in Aims 2 and 3. In Aim 2, the investigators will analyze the location of calls to identify geographic areas with delayed responses for patients with higher severity of illness. As part of their quality assurance/quality improvement practices, Aman Foundation routinely collects location data from GPS devices in their ambulances for each call. Based on the analyses in Aim 2, in Aim 3 the investigators will position ambulances where there are clusters of delayed ambulance calls for high acuity patients to improve response times. This period will be compared with a previous, control period and will be analyzed to identify possible new clusters.

DETAILED DESCRIPTION:
The list of the top causes of death and lost disability-adjusted life-years (DALYs) globally includes many conditions that initially present in the emergency setting. These top causes include lower respiratory infections, ischemic heart disease, and acute injury. The morbidity and mortality that result from these causes can be minimized with emergency treatment. A key element to reducing morbidity and mortality from acute illnesses is the time of patient transport to a medical facility, which has been most clearly demonstrated for acute injury.

Low- and middle-income countries (LMICs) shoulder a disproportionate burden from acute illnesses, yet it has also been demonstrated that reduced transport times to a hospital decrease the odds of mortality in trauma patients in LMICs. A lack of equipment, poorly developed infrastructure, and long distances have been reported as key barriers in the provision of emergency care. Pakistan is one such LMIC that is burdened by many of these challenges in prehospital care. Emergency medical systems (EMS) have only recently been established in Pakistan, and prior to the last several years, patients were routinely transported to healthcare facilities by relatives, bystanders, or by basic patient transport. Where formal patient transport is available, transport times are often prolonged by distance, traffic congestion, and a lack of public cooperation.

Geographic information systems (GIS) are an analytic method that may serve as a key tool in decreasing the time of transporting acutely ill patients to life-saving medical care. GIS, which links geographic information to public health data, has been used in simulations to decrease ambulance response times and been shown to decrease response times in industrialized countries. However, this has not been replicated in other highly developed countries and has never been demonstrated in an LMIC.

The investigators hypothesize that that spatial analysis of the location data of ambulance calls can improve prehospital care provided by Aman Health Care Services in Karachi, Pakistan by decreasing ambulance response times for high acuity patients.

Aim 1: Develop a conceptual framework for prehospital care in LMICs. As no such framework currently exists in the literature, the investigators will develop a conceptual framework to anchor this project in Aims 2 and 3. The framework will be developed after a consideration of other related health systems frameworks in the literature. The investigators will also consult with experts in the field and with the partners in Karachi to comment on how the framework can be improved.

Aim 2: Analyze the location of calls to identify geographic areas with longer calls and higher severity of illness. Using GIS and spatial analysis, the investigators will analyze Aman Ambulance's existing data on ambulance calls to find areas of Karachi that routinely have long response times.

Aim 3: Position ambulances where there are clusters of delayed ambulance calls for high acuity patients to improve response times. Over a six-month period, ambulances will be repositioned in and around clusters of delays to improve response times. This period will be compared with the same calendar period in the previous year using a logistic regression analysis to determine if there is a decrease in delayed ambulance responses. Spatial analyses will also be performed on data from the intervention period to assess for the presence of clusters of delays.

This study has the potential to use a sustainable method of analyzing routinely collected data on ambulance calls to shorten the time that patients with acute illnesses receive appropriate medical care in Pakistan, a setting in which there are substantial infrastructure and human resource challenges.

ELIGIBILITY:
Inclusion Criteria:

* Aman Foundation uses The Medical Priority Dispatch System (MPDS), a commonly used five-tier triage system that includes the following categories (from least to most acute) "alpha," "bravo," "charlie," "delta," and "echo." For the analyses in Aim 2 and Aim 3, we will only examine calls for "delta" and "echo" patients.

Exclusion Criteria:

* Ambulance calls for transport of patients from one healthcare facility to another or calls in which the patient refused transport will be excluded from the analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients in Karachi, Pakistan who call Aman Foundation and request an ambulance.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Ambulance Response Time | 18 months
  Time from when a call comes to the call center to the time the ambulance arrives at the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Kiemanh Pham, MD, MPH, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Aman Foundation, Karachi, Pakistan